CLINICAL TRIAL: NCT01678807
Title: Safety Study of MK-8237 Treatment in House-Dust-Mite Allergic Adolescents (Protocol 008)
Brief Title: Safety Study of MK-8237 Treatment in House-Dust-Mite Allergic Adolescents (MK-8237-008)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ALK-Abelló A/S (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8237-008; MK-8237-008 (Other: Merck Protocol Number)
Record Dates: First submitted 2012-08-31; First posted 2012-09-05 (Estimated); Results first posted 2017-02-13 (Actual); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: Rhinitis, Allergic, Perennial; Rhinitis, Allergic, Nonseasonal
MeSH Terms: conditions — Rhinitis, Allergic, Perennial

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- MK-8237 6 DU (Experimental): MK-8237 6 DU rapidly dissolving tablet administered sublingually once daily for 28 days
  Interventions: Biological: MK-8237 6 DU
- MK-8237 12 DU (Experimental): MK-8237 12 DU rapidly dissolving tablet administered sublingually once daily for 28 days
  Interventions: Biological: MK-8237 12 DU
- Placebo (Placebo Comparator): Placebo rapidly dissolving tablet administered sublingually once daily for 28 days
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: MK-8237 6 DU
  Other Names: SCH 900237
  Arms: MK-8237 6 DU
Biological: MK-8237 12 DU
  Other Names: SCH 900237
  Arms: MK-8237 12 DU
Biological: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety of two doses (6 Development Units [DU] and 12 DU) of MK-8237 sublingual tablets compared to Placebo in adolescents with house dust mite-induced allergic rhinitis/rhinoconjunctivitis. The primary hypothesis is that at least one dose of MK-8237 sublingual tablet is safe and well-tolerated in adolescents with house dust mite-induced allergic rhinitis/rhinoconjunctivitis.

ELIGIBILITY:
Inclusion Criteria:

* History of physician-diagnosed allergic rhinitis/rhinoconjunctivitis to house dust of at least 6 months duration (with or without asthma)
* History of controlled asthma for the prior 1 month if participant has asthma, defined by not exceeding 2 days of symptoms per week; not more than 2 days of albuterol/short acting beta-agonist [SABA] use per week; and not wakening more than twice a month at night due to asthma symptoms
* Agrees to remain abstinent or use (or have their partner use) 2 acceptable methods of birth control from screening and through the duration of the study

Exclusion Criteria:

* Unable to meet medication washout requirements
* History of chronic urticaria and/or chronic angioedema within prior 2 years
* History of anaphylaxis with cardiorespiratory symptoms with prior immunotherapy due to an unknown cause or to an inhalant allergen
* Unstable, uncontrolled or severe asthma, or has experienced a life-threatening asthma attack or an occurrence of any clinical deterioration of asthma that resulted in emergency treatment, hospitalization due to asthma, or treatment with systemic corticosteroids (but allowing SABAs) at any time within prior 3 months
* History of chronic sinusitis during within prior 2 years
* Pregnant or breast-feeding, or expecting to conceive within the projected duration of the study
* Known history of allergy, hypersensitivity or intolerance to investigational medicinal products except for Dermatophagoides pteronyssinus (D. pteronyssinus) and/or Dermatophagoides farina (D. farina) or self-injectable epinephrine
* Business or personal relationship with investigational site personnel or Sponsor who is directly involved with the conduct of the trial

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 195 (Actual)
Dates: Start 2012-10; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Maloney J, Prenner BM, Bernstein DI, Lu S, Gawchik S, Berman G, Kaur A, Li Z, Nolte H. Safety of house dust mite sublingual immunotherapy standardized quality tablet in children allergic to house dust mites. Ann Allergy Asthma Immunol. 2016 Jan;116(1):59-65. doi: 10.1016/j.anai.2015.10.024. Epub 2015 Nov 6. PMID 26553448
- [Derived] Fortescue R, Kew KM, Leung MST. Sublingual immunotherapy for asthma. Cochrane Database Syst Rev. 2020 Sep 14;9(9):CD011293. doi: 10.1002/14651858.CD011293.pub3. PMID 32926419

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants must have had a clinical history of allergic rhinitis/rhinoconjunctivitis (with or without asthma) to house dust of 6 months duration or more and had a positive skin prick test response to Dermatophagoides pteronyssinus or Dermatophagoides farina at the screening visit. Other inclusion and exclusion criteria applied.
Groups:
- MK-8237 12 Development Units (DU): Participants received MK-8237 12 DU rapidly dissolving tablet administered sublingually once daily (q.d.) for 28 days
- MK-8237 6 DU: Participants received MK-8237 6 DU rapidly dissolving tablet administered sublingually q.d. for 28 days
- Placebo: Participants received a rapidly dissolving placebo tablet administered sublingually q.d. for 28 days
Period: Overall Study
Arm/Group | MK-8237 12 Development Units (DU) | MK-8237 6 DU | Placebo
Started | 65 | 65 | 65
Completed | 61 | 60 | 65
Not Completed | 4 | 5 | 0
Not completed — Adverse Event | 4 | 4 | 0
Not completed — Withdrawn by Parent/Guardian | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- MK-8237 12 DU: Participants received MK-8237 12 DU rapidly dissolving tablet administered sublingually once daily (q.d.) for 28 days
- Total: Total of all reporting groups
Arm/Group | MK-8237 12 DU | MK-8237 6 DU | Placebo | Total
Number analyzed (Participants) | 65 | 65 | 65 | 195
Age, Continuous [Mean (Standard Deviation); unit: Years] | 14.5 (1.6) | 14.5 (1.7) | 14.3 (1.8) | 14.4 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 27 | 21 | 73
  Male | 40 | 38 | 44 | 122

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experienced At Least One Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product/protocol-specified procedure, whether or not considered related to the medicinal product/protocol-specified procedure. Any worsening of a preexisting condition temporally associated with the use of the product was also an AE. A serious adverse event (SAE) was an AE that resulted in death, was life threatening, resulted in persistent or significant disability/incapacity, resulted in or prolonged an existing inpatient hospitalization, was a congenital anomaly/birth defect, was a cancer, was associated with an overdose, was another important medical event.
Time Frame: From first dose to last dose of treatment plus 2 weeks of follow-up, up to 42 days
Population: All randomized participants who receive at least one dose of study treatment
Measure: Number; unit: Percentage of participants
Arm/Group | MK-8237 12 DU | MK-8237 6 DU | Placebo
Number analyzed (Participants) | 65 | 65 | 65
Percentage of participants | 56.9 | 53.8 | 43.1
Statistical Analysis 1: Comparison: MK-8237 12 DU vs Placebo; Test type: Superiority or Other; Percent Difference = 13.8, 95% CI 2-sided [-3.4 to 30.3] — Estimate based on Miettinen & Nurminen method stratified by asthma status
Statistical Analysis 2: Comparison: MK-8237 6 DU vs Placebo; Test type: Superiority or Other; Percent Difference = 10.8, 95% CI 2-sided [-6.4 to 27.4] — Estimate based on Miettinen & Nurminen method stratified by asthma status

2. Primary Outcome: Percentage of Participants Who Discontinued Study Drug Due to an Adverse Event
Description: The percentage of participants who had study treatment stopped due to an AE. Discontinuations were reported for all randomized participants who received ≥1 dose of study treatment.
Time Frame: From first dose to last dose of treatment, up to 28 days
Population: All randomized participants who receive at least one dose of study treatment
Measure: Number; unit: Percentage of participants
Arm/Group | MK-8237 12 DU | MK-8237 6 DU | Placebo
Number analyzed (Participants) | 65 | 65 | 65
Percentage of participants | 6.2 | 6.2 | 0
Statistical Analysis 1: Comparison: MK-8237 12 DU vs Placebo; Test type: Superiority or Other; Percent Difference = 6.2, 95% CI 2-sided [0.4 to 14.8] — Estimate based on Miettinen & Nurminen method stratified by asthma status
Statistical Analysis 2: Comparison: MK-8237 6 DU vs Placebo; Test type: Superiority or Other; Percent Difference = 6.2, 95% CI 2-sided [0.4 to 14.8] — Estimate based on Miettinen & Nurminen method stratified by asthma status

ADVERSE EVENTS:
Time Frame: From first dose to last dose of treatment plus 2 weeks of follow-up, up to 42 days
Description: Adverse events for all randomized participants who receive at least one dose of study treatment
Arm/Group | MK-8237 12 DU | MK-8237 6 DU | Placebo
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/65 | 0/65
Other Adverse Events (participants affected / at risk) | 29/65 | 27/65 | 12/65
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-8237 12 DU (N=65) | MK-8237 6 DU (N=65) | Placebo (N=65)
Ear pruritus (Ear and labyrinth disorders) | 1 (1) | 5 (22) | 1 (2)
Lip swelling (Gastrointestinal disorders) | 7 (10) | 3 (5) | 0 (0)
Oral pruritus (Gastrointestinal disorders) | 11 (31) | 11 (40) | 5 (11)
Paraesthesia oral (Gastrointestinal disorders) | 5 (13) | 6 (11) | 1 (1)
Tongue pruritus (Gastrointestinal disorders) | 6 (14) | 9 (19) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 5 (5) | 2 (2)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 13 (36) | 12 (24) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor has the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results.